CLINICAL TRIAL: NCT03056703
Title: An Open Label, Randomized, Two-Way Crossover Trial to Assess the Bioequivalence of a Single Oral Dose of a 1000 mg Fast Release Aspirin Tablet Versus Two 500 mg Fast Release Aspirin Tablets in Healthy Male and Female Subjects
Brief Title: Bioequivalence of Single Dose Fast Release Aspirin (1000 mg) Tablet Versus Single Dose of Two 500 mg Fast Release Aspirin Tablets
Acronym: Mille
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 16645
Record Dates: First submitted 2017-02-15; First posted 2017-02-17 (Actual); Last update posted 2017-02-17 (Actual); Status verified 2017-02

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acetylsalicylic acid [1000mg] (Experimental)
  Interventions: Drug: Acetylsalicylic acid (Aspirin, BAY1019036)
- Acetylsalicylic acid [500mg] (Active Comparator)
  Interventions: Drug: Acetylsalicylic acid (Aspirin, BAY1019036)

INTERVENTIONS:
Drug: Acetylsalicylic acid (Aspirin, BAY1019036) — One Fast Release Tablet containing 1000 mg acetylsalicylic acid
  Arms: Acetylsalicylic acid [1000mg]
Drug: Acetylsalicylic acid (Aspirin, BAY1019036) — Two Fast Release Tablets containing 500 mg acetylsalicylic acid each
  Arms: Acetylsalicylic acid [500mg]

SUMMARY:
The primary objective of this study is to compare the bioavailability of a single dose of a new 1000 mg fast release ASA (acetylsalicylic acid) tablet with that of two tablets of a commercially available 500 mg fast release tablet and to test for bioequivalence of the new versus the commercial product in healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy ambulatory male and female subjects 18 to 55 years of age, inclusive
* Body Mass Index (BMI) of approximately 18.5 to 30.0 kg/m2, and a total body weight >50 kg (110 lbs)
* Results of screening and clinical laboratory tests are within normal limits or considered not clinically significant by the Principal Investigator or Sponsor
* Female subjects of childbearing potential must be using a medically acceptable form of birth control for at least 1 month prior to screening (3 months on oral contraceptives), e.g., oral or patch contraceptives, intrauterine device, intramuscular injection or double-barrier and have a negative pregnancy test at Screening and on Day 0 of each treatment period. Female subjects of nonchildbearing potential must be amenorrheic for at least 2 years or had a hysterectomy and/or bilateral oophorectomy.
* Provide a personally signed and dated informed consent prior to inclusion in the trial indicating that the subject has been informed of all pertinent aspects of the trial.

Exclusion Criteria:

* History of hypersensitivity to acetylsalicylic acid (ASA), naproxen sodium, acetaminophen, other non-steroidal anti-inflammatory drugs (NSAIDs), and similar pharmacological agents or components of the products
* History of gastrointestinal bleeding or perforation, including bleeding related to previous NSAID therapy. Active, or history of recurrent peptic ulcer/hemorrhage (two or more distinct episodes of proven ulceration or bleeding).
* Have taken ASA, ASA-containing products, acetaminophen or any other NSAID (OTC or prescription) seven days prior to dosing or during the Treatment Periods, other than study product
* Loss of blood in excess of 500 mL within 56 days of the first dose of trial treatment (e.g., donation, plasmapheresis, or injury)
* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic disease, or malignancies
* Positive alcohol or drug screen at Screening or on Day 0 of Treatment Periods 1 or 2
* Females who are pregnant or lactating
* Consumption of xanthine-containing food and beverages within 24 h before investigational medicinal product (IMP) administration during Treatment Periods 1 and 2; or not willing to abstain from any xanthine containing food and beverages during the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Estimated)
Dates: Start 2014-02; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
AUC0-inf (area under plasma concentration versus time curve) for ASA (acetylsalicylic acid) | baseline (pre-dose) and 5, 7.5, 10, 12.5, 15, 17.5, 20, 22.5, 25, 27.5, 30, 35, 40, 45, 50, 55 minutes and 1. 1.25, 1.5, 2, 3, 4, 5, 6, 8, 12, and 24 hours post-dose
AUC0-t for ASA | baseline (pre-dose) and 5, 7.5, 10, 12.5, 15, 17.5, 20, 22.5, 25, 27.5, 30, 35, 40, 45, 50, 55 minutes and 1. 1.25, 1.5, 2, 3, 4, 5, 6, 8, 12, and 24 hours post-dose
Cmax (maximum plasma concentration) for ASA | baseline (pre-dose) and 5, 7.5, 10, 12.5, 15, 17.5, 20, 22.5, 25, 27.5, 30, 35, 40, 45, 50, 55 minutes and 1. 1.25, 1.5, 2, 3, 4, 5, 6, 8, 12, and 24 hours post-dose

SECONDARY OUTCOMES:
AUC0-inf for SA (salicylic acid) | baseline (pre-dose) and 5, 7.5, 10, 12.5, 15, 17.5, 20, 22.5, 25, 27.5, 30, 35, 40, 45, 50, 55 minutes and 1. 1.25, 1.5, 2, 3, 4, 5, 6, 8, 12, and 24 hours post-dose
AUC0-t for SA | baseline (pre-dose) and 5, 7.5, 10, 12.5, 15, 17.5, 20, 22.5, 25, 27.5, 30, 35, 40, 45, 50, 55 minutes and 1. 1.25, 1.5, 2, 3, 4, 5, 6, 8, 12, and 24 hours post-dose
Cmax for SA | baseline (pre-dose) and 5, 7.5, 10, 12.5, 15, 17.5, 20, 22.5, 25, 27.5, 30, 35, 40, 45, 50, 55 minutes and 1. 1.25, 1.5, 2, 3, 4, 5, 6, 8, 12, and 24 hours post-dose
t1/2 for ASA and SA | baseline (pre-dose) and 5, 7.5, 10, 12.5, 15, 17.5, 20, 22.5, 25, 27.5, 30, 35, 40, 45, 50, 55 minutes and 1. 1.25, 1.5, 2, 3, 4, 5, 6, 8, 12, and 24 hours post-dose
tmax for ASA and SA | baseline (pre-dose) and 5, 7.5, 10, 12.5, 15, 17.5, 20, 22.5, 25, 27.5, 30, 35, 40, 45, 50, 55 minutes and 1. 1.25, 1.5, 2, 3, 4, 5, 6, 8, 12, and 24 hours post-dose
Lambda(z) (terminal rate constant) for ASA and SA | baseline (pre-dose) and 5, 7.5, 10, 12.5, 15, 17.5, 20, 22.5, 25, 27.5, 30, 35, 40, 45, 50, 55 minutes and 1. 1.25, 1.5, 2, 3, 4, 5, 6, 8, 12, and 24 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Hackensack, New Jersey, United States